CLINICAL TRIAL: NCT03493867
Title: Verification Protocol for The Cloud DX Vitaliti™ Continuous Vital Sign Monitor (CVSM): Non-invasive Blood Pressure Component for Clinical Use and Self Measurement According to the American Safety in Medical Technology and the IEEE
Brief Title: Verification of The Cloud DX Vitaliti™ Continuous Vital Sign Monitor (CVSM): Non-invasive Blood Pressure Component
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Collaborators: Federal Economic Development Agency for Southern Ontario (FedDev Ontario) (Other)
Responsible Party: Principal Investigator, Mike McGillion, Associate Professor and Assistant Dean, Population Health Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STP-VIT-002
Record Dates: First submitted 2018-03-16; First posted 2018-04-11 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Blood Pressure
Keywords: Non-invasive blood pressure monitoring; Wearable device; Medical device verification study

STUDY DESIGN:
Intervention Model Description: Vitaliti Continuous Vital Sign Monitoring Device - Version 2.0
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vitaliti (Other): The subject's blood pressure will be simultaneously determined and recorded using the invasive arterial line blood pressure reading and the test Vitaliti device readings.
  Interventions: Device: Vitaliti

INTERVENTIONS:
Device: Vitaliti — Measurements recorded by the Vitaliti device will be compared to the recordings from the arterial catheter.

SUMMARY:
The purpose of this study is the verification of Cloud-DX Vitaliti™ Continuous Automated Non-Invasive Blood Pressure Monitor for Clinical Use and Self Measurement according to standards laid out by IEEE Std 1708 and AAMI-ISO 81060-2.

DETAILED DESCRIPTION:
Several automated vital sign measurement systems have been developed recently; however, non-invasive continuous blood pressure monitoring continues to be a major limitation. To circumvent the limitations of current systems of interval hemodynamic measurement and increasing demands on health care providers, a non-invasive automated continuous vital sign monitor that can integrate into hospital early warning systems and warn health care providers of deteriorating vital sign parameters would be of significant value and a major advance for current hospital monitoring systems.

Cloud-DX Vitaliti™ is a new low profile automated vital sign monitor, which includes a continuous non-invasive blood pressure measurement system. Additional parameters are also measured. Paired with companion software from cloud based computing, Vitaliti™ features a user friendly interface, onboard radios for communication with smartphones/tablets/personal computers, and several sensors.

Cloud-DX Vitaliti™ has undergone preliminary testing and is now ready for verification to achieve compliance with AAMI/ISO and IEEE standards of medical grade device. At the Hamilton General Hospital (HGH), Cardiac Surgical Intensive Care Unit (CICU) and Vascular Surgical Step Down Units, arterial catheters are standard of care and performed on most patients for variable periods of post-operative recovery. Within this setting, the IEEE Std 1708 and AAMI-ISO 81060-2 would be fully met. Furthermore, the cardiovascular surgical caseloads at HGH would provide sufficient test subjects to validate VitalitiTM in a timely fashion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age;
2. Patient has undergone major cardiac or vascular surgery and has been admitted post-op to the cardiac surgical intensive care unit (CICU) or vascular surgery step down unit with an arterial line in place

Exclusion Criteria:

1. Patients < 18 years of age;
2. Pregnant;
3. Current arrhythmia
4. Blood pressure outside of test range for phase (refer to table 1)
5. Allergy to device contact adhesive (e.g. ECG leads)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2019-11-06 (Actual); Study Completion 2019-11-06 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 30 minutes
  Determining the accuracy of non-invasive blood pressure measurement compared to invasive blood pressure. A detailed analysis will be conducted on the invasive blood pressure to verify accuracy as defined in the ISO 81060-2 Standard.

CONTACTS AND LOCATIONS:
Overall Officials: Michael McGillion, RN, PhD, Principal Investigator — School of Nursing, Faculty of Health Sciences, McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided
The data which will be collected is only valid for the verification of this particular device.

REFERENCES:
- [Derived] McGillion MH, Dvirnik N, Yang S, Belley-Cote E, Lamy A, Whitlock R, Marcucci M, Borges FK, Duceppe E, Ouellette C, Bird M, Carroll SL, Conen D, Tarride JE, Harsha P, Scott T, Good A, Gregus K, Sanchez K, Benoit P, Owen J, Harvey V, Peter E, Petch J, Vincent J, Graham M, Devereaux PJ. Continuous Noninvasive Remote Automated Blood Pressure Monitoring With Novel Wearable Technology: A Preliminary Validation Study. JMIR Mhealth Uhealth. 2022 Feb 28;10(2):e24916. doi: 10.2196/24916. PMID 34876396